CLINICAL TRIAL: NCT03918915
Title: A Multicenter, Randomized, Double-masked, Vehicle-controlled Study to Assess the Safety and Efficacy of SYD-101 Ophthalmic Solution for the Treatment of Myopia in Children
Brief Title: The Safety and Efficacy of SYD-101 in Children With Myopia
Acronym: STAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sydnexis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYD-101-001
Record Dates: First submitted 2019-04-12; First posted 2019-04-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Nearsightedness; Near Sightedness; Near-sightedness
Keywords: Children; Myopia
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SYD-101 0.01% (Experimental): 1 drop in each eye at bedtime. Part 1: participants will be randomized to SYD-101 0.01% Part 2: participants will be re-randomized to SYD-101 0.01% or Vehicle
  Interventions: Drug: SYD-101 0.01%
- SYD-101 0.03% (Experimental): 1 drop in each eye at bedtime. Part 1: participants will be randomized to SYD-101 0.03% Part 2: participants will be re-randomized to SYD-101 0.03% or Vehicle
  Interventions: Drug: SYD-101 0.03%
- Vehicle (Placebo Comparator): 1 drop in each eye at bedtime. Part 1: participants will be randomized to Vehicle Part 2: participants will be re-randomized to SYD-101 0.03%
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: SYD-101 0.01% — Sterile topical ophthalmic solution
  Other Names: atropine sulfate
  Arms: SYD-101 0.01%
Drug: SYD-101 0.03% — Sterile topical ophthalmic solution
  Other Names: atropine sulfate
  Arms: SYD-101 0.03%
Drug: Vehicle — Sterile topical ophthalmic solution without active ingredient
  Other Names: Placebo
  Arms: Vehicle

SUMMARY:
Myopia, or nearsightedness, is the most common eye disorder, often affecting more than 40% of adults in Europe, Asia and the USA. Severe myopia is associated with an increased risk of developing other eye conditions such as glucoma, cataracts and retinal detachment, which may lead to blindness. Early treatment of myopia in children could help slow the condition and minimize the risk of complications later in life. This study investigates the use of SYD-101, an eye solution, in slowing-down the progression of myopia in children.

DETAILED DESCRIPTION:
This will be a 3-arm, multicentered, randomized, double-masked, vehicle-controlled study conducted in 2 parts.

Part 1 is the primary treatment period of 3 years, during which participants will receive 1 of 3 masked medications.

Part 2 is the randomized withdrawal period of 1 year, during which participants originally receiving Vehicle will receive SYD-101, and participants originally receiving SYD-101 will receive either Vehicle or SYD-101.

ELIGIBILITY:
Inclusion Criteria:

* Myopia of 0.5 D (diopters) to 6.00 D (inclusive) in both eyes.
* Astigmatism ≤1.50 D in both eyes.
* Anisometropia ≤1.00 D in both eyes.
* If myopia is ≥0.75 D, participant must be wearing single vision eyeglasses or soft, daily-wear, single-vision contact lenses that meet study investigator's criteria.
* BCVA (best-corrected visual acuity) Snellen equivalent of 20/32 or better.

Exclusion Criteria:

* Participants with a history or current evidence of a medical condition predisposing them to degenerative myopia (e.g. Marfan syndrome, Stickler syndrome), or a condition that may affect visual function or development (e.g. diabetes mellitus, chromosome anomaly).
* Current use of a monoamine oxidase inhibitor.
* Evidence of any ocular inflammation or infection in either eye, including blepharitis, conjunctivitis, keratitis, and scleritis.
* Past, present or future plans to use orthokeratology (orthoK), rigid gas-permeable, bifocal, progressive-addition, multi-focal, or other lenses to reduce myopia progression; or the use of atropine, pirenzepine or other anti-muscarinic agent for myopia.
* History or evidence of ocular surgery or planned future ocular surgery in either eye.

Other protocol-defined inclusion/exclusion criteria could apply.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 852 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Myopic progression >0.75 D (diopters) | Month 36
  Proportion of participants with confirmed myopic progression >0.75 D (diopters), based on SE (spherical equivalent) as measured by cycloplegic autorefraction

SECONDARY OUTCOMES:
Mean annual myopic progression | Month 36
  Mean annual progression rate of myopia measured in diopters: Spherical Equivalent (SE) as measured by cycloplegic autorefraction.
Proportion of participants with annual myopia progression rate <=0.50 D/year | Through Month 36
  Mean annual progression rate of myopia
Proportion of participants with annual myopia progression rate <=0.25 D/year | Through Month 36
  Mean annual progression rate of myopia
Proportion of participants with annual myopia progression rate > 0.50 D/year | Month 36
  Mean annual progression rate of myopia
Time to progression of myopia >0.75 D (diopters) | Up to 36 months (from date of randomization until date myopia progresses >0.75 D)
  Progression of myopia measured as Spherical Equivalent (SE) via cycloplegic autorefraction.
Mean change from baseline in axial length (subset only) | Baseline to Month 36
  Measured by cycloplegic biometry

CONTACTS AND LOCATIONS:
Locations (47):
- United States (41):
  - Site 143, Irwindale, California
  - Site 144, Pasadena, California
  - Site 148, San Diego, California
  - Site 104, San Diego, California
  - Site 110, Santa Barbara, California
  - Site 133, Sunnyvale, California
  - Site 130, Colorado Springs, Colorado
  - Site 100, Fort Collins, Colorado
  - Site 102, Danbury, Connecticut
  - Site 150, Waterbury, Connecticut
  - Site 122, Fort Lauderdale, Florida
  - Site 109, Jupiter, Florida
  - Site 119, Sweetwater, Florida
  - Site 120, Tamarac, Florida
  - Site 124, Marietta, Georgia
  - Site 116, Chicago, Illinois
  - Site 106, Wilmette, Illinois
  - Site 135, Indianapolis, Indiana
  - Site 131, Munster, Indiana
  - Site 137, Pittsburg, Kansas
  - Site 138, Bangor, Maine
  - Site 123, Boston, Massachusetts
  - Site 114, Washington, Missouri
  - Site 132, Henderson, Nevada
  - Site 139, Albuquerque, New Mexico
  - Site 127, Buffalo, New York
  - Site 117, Chapel Hill, North Carolina
  - Site 121, Raleigh, North Carolina
  - Site 105, Fargo, North Dakota
  - Site 111, Medford, Oregon
  - Site 147, Tigard, Oregon
  - Sie 136, Bala-Cynwyd, Pennsylvania
  - Site 128, Cranberry Township, Pennsylvania
  - Site 108, Charleston, South Carolina
  - Site 126, Lakeway, Texas
  - Site 142, San Antonio, Texas
  - Site 101, San Antonio, Texas
  - Site 115, The Woodlands, Texas
  - Site 149, Ogden, Utah
  - Site 140, Ogden, Utah
  - Site 113, Virginia Beach, Virginia
- Austria (3):
  - Site 204, Graz, Styria
  - Site 203, Linz, Upper Austria
  - Site 205, Vienna
- Slovakia (3):
  - Site 202, Bratislava
  - Site 201, Trebišov
  - Site 200, Trenčín

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson P, Widder K, Cheetham J, Kirkeby L. Methods and baseline of a large, multicenter, phase 3 study with low-dose atropine (SYD-101) for the treatment of myopia progression in over 800 children (STAR Study). Invest Ophthalmol Vis Sci. 2025; 66(8), 2825
- [Background] Cheetham JK, Gieschen L, Kirkeby L, Widder K, Johnson P. The natural history of myopia progression in a large diverse pediatric population. Invest Ophthalmol Vis Sci. 2025; 66(8), 2824
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls

DOCUMENTS (2):
  • Study Protocol (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT03918915/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT03918915/SAP_001.pdf